CLINICAL TRIAL: NCT01225146
Title: A Phase I Open Label Study of the Safety, Tolerability and Efficacy of 2.0 mg Ranibizumab in Subjects With Ischemic Central Retinal Vein Occlusion (RAVE2)
Brief Title: Study of 2.0 mg Ranibizumab in Subjects With Ischemic Central Retinal Vein Occlusion (RAVE2)
Acronym: RAVE2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The collaborator, Genentech, stopped supplying the study drug to the site.
Sponsor: David M. Brown, M.D. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David M. Brown, M.D., Director of Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4820s
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-05

CONDITIONS: Ischemia; Retinal Vein Occlusion; Pathologic Processes; Retinal Diseases; Eye Diseases
Keywords: Ischemic; Central; Retinal; Vein; Occlusion; Ranibizumab; Lucentis; CRVO; ISCRVO
MeSH Terms: conditions — Ischemia; Retinal Vein Occlusion; Pathologic Processes; Retinal Diseases; Eye Diseases; Bites and Stings | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Experienced (Cohort 1 (Active Comparator): Previously treated with 6 or more intravitreal ranibizumab with persistent edema followed in RAVE 1 (FVF3348s).
  Cohort 1 patients will receive 1 dose of ranibizumab 2.0 mg, followed by PRN based on pre-defined retreatment criteria
  Interventions: Drug: ranibizumab
- Treatment Naive (Cohort 2) (Active Comparator): Treatment naïve. Cohort 2 patients will receive 6 doses of ranibizumab 2.0 mg, followed by PRN based on pre-defined re-treatment criteria.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Ranibizumab is formulated as a sterile solution aseptically filled in a sterile 3-mL stoppered glass vial. Each vial contains 0.5 mL of 40 mg/mL (2.0-mg dose level) ranibizumab aqueous solution.
  Other Names: Lucentis

SUMMARY:
The RAVE 2 trial is a phase I, open label, 12-month trial of intravitreal ranibizumab 2.0 mg in patients with ischemic CRVO who have been either previously treated with ranibizumab or treatment naïve.

DETAILED DESCRIPTION:
The most devastating complication of ischemic CRVO is the development of anterior segment neovascularization and the resulting morbidity from neovascular glaucoma. This complication appears to be directly correlated with intraocular VEGF levels. Currently there is no proven treatment to decrease the formation of rubeosis. Current management of the disease consists of pan-retinal photocoagulation once significant anterior segment neovascularization becomes manifest. This treatment destroys peripheral retina (with peripheral retinal field) and presumably works by eventually lowering ocular VEGF levels which causes secondary regression of rubeosis.

As ranibizumab blocks VEGF, this treatment when delivered intraocularly may prevent neo-vascular glaucoma while preserving peripheral visual fields in this patient population.

A higher dose of ranibizumab may allow for both a longer duration of treatment effect and potentially more efficacy leading to better outcomes for patients that are somewhat treatment resistant and need continual therapy. Nonclinical and early clinical data indicate that higher doses of ranibizumab up to and including 2.0 mg are safe and tolerated by patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  * Ability to provide written informed consent and comply with study assessments for the full duration of the study
  * Age > 18 years
  * For patients previously treated with ITV ranibizumab (Cohort 1):
  * 6 or more intravitreal injections of ranibizumab with presence of persistent edema after a minimum of 6 ranibizumab injections followed in RAVE 1.
  * For treatment naïve (Cohort 2):
  * Ischemic CRVO within 3 months of enrollment as per the following inclusion criteria

Three of the following clinical tests must be present to demonstrate ischemic CRVO:

* VA 20/200 or worse
* RAPD 0.9 LU or worse
* Loss of 1-2e isopter on Goldmann Visual field (Kwon et al. 2001)
* ERG demonstrating b wave amplitude less than 60% of A wave
* Capillary nonperfusion greater than 50 DA

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  * IOP over 30 mm Hg
  * Any previous retinal laser photocoagulation to the study eye in treatment naive
  * Any previous intravitreal injection in study eye (triamcinolone or other) in treatment naive
  * Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery)
  * Intracapsular cataract extraction (posterior capsule needs to be present)
  * Previous history of retinal detachment in study eye
  * Any previous radiation treatments to head/ neck
  * Inability to assess iris neovascularization (corneal opacity precluding gonioscopy)
  * Significant cardiovascular disease or cancer that would prevent follow-up visits or completion of the 12 month study
  * Significant diabetic retinopathy in the fellow eye (diabetic macular edema, proliferative diabetic retinopathy, or high-risk non-proliferative diabetic retinopathy)
  * Pregnancy (positive pregnancy test)
  * Participation in another simultaneous medical investigator or trial
  * Ocular disorders in the study eye that may confound interpretation of study results, including retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., DME AMD, ocular histoplasmosis, or pathologic myopia)
  * Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period
  * Aphakia or absence of the posterior capsule in the study eye
  * Previous violation of the posterior capsule is also excluded unless it occurred as a result of YAG laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
  * History of idiopathic or autoimmune uveitis in either eye
  * Structural damage to the center of the macula in the study eye preexisting to CRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s)
  * Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
  * Ocular inflammation (including trace or above) in the study eye
  * Infectious blepharitis, keratitis, scleritis, or conjunctivitis (in either eye) or current treatment for serious systemic infection
  * Spherical equivalent of the refractive error in the study eye of more than -8 diopters myopia (For patients who have had refractive or cataract surgery in the study eye, pre-operative spherical equivalent refractive error of more than -8 diopters myopia is not allowed)

Systemic Conditions

* Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period
* Uncontrolled diabetes mellitus
* Renal failure requiring dialysis or renal transplant
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* History of other disease, metabolic dysfunction, physical examination finding, or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications

Other

* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow up procedures
* History of allergy to humanized antibodies or any component of the ranibizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Wykoff, MD, PhD, Principal Investigator — Retina Consultants Houston
Locations (1):
- Retina Consultants of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wykoff CC, Brown DM, Croft DE, Major JC Jr, Wong TP. Progressive retinal nonperfusion in ischemic central retinal vein occlusion. Retina. 2015 Jan;35(1):43-7. doi: 10.1097/IAE.0000000000000277. PMID 25102193

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Experienced (Cohort 1: Previously treated with 6 or more intravitreal ranibizumab with persistent edema followed in RAVE 1 (FVF3348s).
  Cohort 1 patients will receive 1 dose of ranibizumab 2.0 mg, followed by PRN based on pre-defined retreatment criteria
  ranibizumab: Ranibizumab is formulated as a sterile solution aseptically filled in a sterile 3-mL stoppered glass vial. Each vial contains 0.5 mL of 40 mg/mL (2.0-mg dose level) ranibizumab aqueous solution.
Period: Overall Study
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Started | 6 | 2
Completed | 6 | 0
Not Completed | 0 | 2
Not completed — Sponsor discontinued making 2mg drug | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Previously treated with 6 or more intravitreal ranibizumab with persistent edema followed in RAVE 1 (FVF3348s).
  Cohort 1 patients will receive 1 dose of ranibizumab 2.0 mg, followed by PRN based on pre-defined retreatment criteria
  ranibizumab: Ranibizumab is formulated as a sterile solution aseptically filled in a sterile 3-mL stoppered glass vial. Each vial contains 0.5 mL of 40 mg/mL (2.0-mg dose level) ranibizumab aqueous solution.
- Cohort 2: Treatment naïve. Cohort 2 patients will receive 6 doses of ranibizumab 2.0 mg, followed by PRN based on pre-defined re-treatment criteria.
  ranibizumab: Ranibizumab is formulated as a sterile solution aseptically filled in a sterile 3-mL stoppered glass vial. Each vial contains 0.5 mL of 40 mg/mL (2.0-mg dose level) ranibizumab aqueous solution.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 64.7 [47 to 76] | 56.5 [42 to 71] | 62.6 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in logMAR
Description: Mean change from baseline in ETDRS NCVA.
Time Frame: 12 months.
Population: Patients in cohort 2 did not complete the study.
Measure: Mean (Full Range); unit: logMAR
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Number analyzed (Participants) | 6 | 0
logMAR | 0.91 [0.4 to 1.42] |

2. Secondary Outcome: Incidence and Severity of Adverse Events (Ocular and Non-ocular).
Description: Incidence and severity of adverse events (ocular and non-ocular) from baseline through 12 months will be evaluated.
Time Frame: 12 months
Measure: Number; unit: incidents
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Number analyzed (Participants) | 6 | 2
incidents
  Ocular Events | 1 | 0
  Non-Ocular Events | 0 | 0
  Serious Ocular Events | 0 | 0
  Serious Non-Ocular Events | 0 | 0

3. Secondary Outcome: Neovascularization Development
Description: Percent of patients that develop neovascularization of the iris, optic nerve and/or elsewhere.
Time Frame: 12 months
Population: Patients in cohort 2 did not complete the study.
Measure: Number; unit: Percentage of patients
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Number analyzed (Participants) | 6 | 0
Percentage of patients | 0 |

4. Secondary Outcome: Mean Change in Central Foveal Volume
Description: Mean change in Central Foveal Volume on High Resolution OCT
Time Frame: 12 months
Population: Patients in cohort 2 did not complete the study.
Measure: Mean (Full Range); unit: mm^3
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Number analyzed (Participants) | 6 | 0
mm^3 | 0.03 [-0.03 to 0.24] |

5. Secondary Outcome: Changes, by Disc Areas, of Capillary Non-perfusion in the Periphery
Description: Changes, by disc areas, of capillary non-perfusion in the periphery (evaluated by wide-field fluorescein angiography) at 3, 6, 9 and 12 months from baseline.
Time Frame: 12 months
Population: Data for this outcome measure were not collected. The study was terminated because the collaborator, Genentech, stopped production of the study drug (2.0 mg ranibizumab). Analysis of this outcome was therefore deferred and is being rolled over to the WAVE study program (NCT01710839, IND 12246)
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Goldman Visual Field Changes
Description: Goldman Visual Field changes at 6 and 12 months from baseline
Time Frame: 12 months
Population: as for outcome 5
Arm/Group | Treatment Experienced (Cohort 1 | Treatment Naive (Cohort 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Ocular and non-ocular adverse events were documented.
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=2)
Increased cup to disk ratio (Eye disorders) | 1 | 0 — OD

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No